CLINICAL TRIAL: NCT06761092
Title: Nebulized Dexmedetomidine to Reduce Post-Anesthesia Delirium of Sevoflurane in Preschool Children Undergoing Elective Surgery
Brief Title: Nebulized Dexmedetomidine for Post-Anesthesia Delirium in Preschool Children
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Jimmy Wongkar, Medical Doctor, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP.04.03/D.XVII.2.2.2/76407/24
Record Dates: First submitted 2024-12-29; First posted 2025-01-07 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Emergence Delirium; Delirium - Postoperative
Keywords: nebulized; dexmedetomidine; post anesthesia delirium; sevoflurane; preschool
MeSH Terms: conditions — Emergence Delirium | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: pediatric preschool, age 2-6 years old, undergoing elective general surgery
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebulized Dexmedetomidine for Post-Anesthesia Delirium in Preschool Children (Active Comparator): Nebulization with the anesthetic drug dexmedetomidine at a dose of 2 mcg/kg body weight, diluted to 3 ml with 0.9% normal saline, administered before the induction of anesthesia in the reception area.
  After the anesthesia, primary data collection is conducted by recovery room staff who are blinded to the treatment and control groups. Data includes scores or levels of post-anesthesia delirium or agitation assessed using the pediatric anesthesia emergence delirium score (PAED score) at 15, 30, 60, and 120 minutes post-surgery in the recovery room.
  Interventions: Drug: Nebulized Dexmedetomidine for Post-Anesthesia Delirium in Preschool Children
- Nebulized Normal Saline 0.9% for Post-Anesthesia Delirium in Preschool Children (Placebo Comparator): Nebulization with normal saline 0.9% 3ml, administered before the induction of anesthesia in the reception area. After the anesthesia, primary data collection is conducted by recovery room staff who are blinded to the treatment and control groups. Data includes scores or levels of post-anesthesia delirium or agitation assessed using the pediatric anesthesia emergence delirium score (PAED score) at 15, 30, 60, and 120 minutes post-surgery in the recovery room.
  Interventions: Procedure: Nebulized 0.9% Normal Saline

INTERVENTIONS:
Drug: Nebulized Dexmedetomidine for Post-Anesthesia Delirium in Preschool Children — Nebulization with the anesthetic drug dexmedetomidine at a dose of 2 mcg/kg body weight, diluted to 3 ml with 0.9% normal saline, administered before the induction of anesthesia in the reception area.
  After the anesthesia, primary data collection is conducted by recovery room staff who are blinded to the treatment and control groups. Data includes scores or levels of post-anesthesia delirium or agitation assessed using the PAED score at 15, 30, 60, and 120 minutes post-surgery in the recovery room
  Arms: Nebulized Dexmedetomidine for Post-Anesthesia Delirium in Preschool Children
Procedure: Nebulized 0.9% Normal Saline — Nebulization with normal saline 0.9% 3 ml, administered before the induction of anesthesia in the reception area. After the anesthesia, primary data collection is conducted by recovery room staff who are blinded to the treatment and control groups. Data includes scores or levels of post-anesthesia delirium or agitation assessed using the PAED score at 15, 30, 60, and 120 minutes post-surgery in the recovery room
  Arms: Nebulized Normal Saline 0.9% for Post-Anesthesia Delirium in Preschool Children

SUMMARY:
Analyzing the effectiveness of nebulized dexmedetomidine 2 mcg/kg in reducing the incidence of post-anesthesia delirium in preschool children undergoing elective surgery with sevoflurane inhalation general anesthesia.

Researchers will compare nebulized Dexmedetomidine to a placebo (a look-alike substance that contains no drug) to see if the drug can reduce post anesthesia delirium incidence.

DETAILED DESCRIPTION:
participant will : Nebulized with the anesthetic drug dexmedetomidine at a dose of 2 mcg/kg body weight, diluted to 3 ml with 0.9% normal saline, is administered before the induction of anesthesia in the reception area.

After the anesthesia, primary data collection is conducted by recovery room staff who are blinded to the treatment and control groups. Data includes scores or levels of post-anesthesia delirium or agitation assessed using the pediatric anesthesia emergence delirium score (PAED score) in the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 2 to 6 years old.
* Planned general anesthesia using inhalation sevoflurane with endotracheal tube techniques
* Parents agree to participate in the study

Exclusion Criteria:

* Pediatric patients with > ASA II.
* Difficult airway management.
* Emergency surgery.
* Congenital abnormalities of vital organs.
* Malnutrition
* history or diagnosed with mental or cognitive disorders.
* History of upper respiratory infection within 2 weeks before the procedure.
* History of allergy to dexmedetomidine.
* Surgery duration estimation exceeding 180 minutes.
* Parents refuse to participate in the study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-02-07 (Estimated); Study Completion 2025-02-13 (Estimated)

PRIMARY OUTCOMES:
reduce post anesthesia delirium incidence | 120 minutes (after extubation till discharge from recovery room)
  After the anesthesia, primary data collection is conducted by recovery room staff who are blinded to the treatment and control groups. Data includes scores or levels of post-anesthesia delirium or agitation assessed using the PAED score at 15, 30, 60, and 120 minutes post-surgery in the recovery room.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive Therapy Udayana University, Denpasar, Bali, Indonesia